CLINICAL TRIAL: NCT02925728
Title: Nutritional Intake of "Finger-food" on Elderly People in Seniors's Resident
Acronym: FIFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHD052-16
Record Dates: First submitted 2016-09-27; First posted 2016-10-06 (Estimated); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-03

CONDITIONS: Nutritive Value
Keywords: Finger-Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition with Finger-Food (Experimental): Nutrition with Finger-Food
  Interventions: Other: Finger-Food
- Nutrition without Finger-Food (Active Comparator): Nutrition without Finger-Food
  Interventions: Other: Without Finger-Food

INTERVENTIONS:
Other: Finger-Food — Finger-Food at lunch and having diner
  Arms: Nutrition with Finger-Food
Other: Without Finger-Food — Without finger-food
  Arms: Nutrition without Finger-Food

SUMMARY:
The undernourishment and the prevention of its risk at the elderly person in seniors's resident represent a major issue in public health. The diagnosis of undernourishment and its risk are systematically recommended in these structures where the nutrition of these people is a problem because often inappropriate for their capacities of prehension and consequently for their nutritional needs. One of the solutions to remedy can be found in the " finger-food ".

The study FIFO ("Finger-Food") suggests verifying the hypothesis which the finger-food would allow to increase the nutritional intake of the resident who have disorders of the prehension and\or requiring a nutritional stimulation and\or require an help to the preparation of the meal.

ELIGIBILITY:
Inclusion Criteria:

* Residents institutionalized in seniors's resident for 3 months at least
* Residents in disability to feed single-handedly because of cognitive and/or physical disorders
* Having at least use of a hand
* Do not opposing the participation in the study or information and not opposition of the family / close to confidence / legal guardian in case of resident in incapacity to understand (senility, insanity)

Exclusion Criteria:

* Confined to bed
* Specific diets (without residue, allergen, …)
* Enteral nutrition
* Absence motricity of 2 hands

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Departemental Vendée, La Roche-sur-Yon, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nutrition With Finger-Food | Nutrition Without Finger-Food
Started | 22 | 25
Completed | 17 | 20
Not Completed | 5 | 5
Not completed — Death | 3 | 5
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Exclusion of 4 patients from the intention-to-treat analysis (for whom at least one post-randomisation efficacy endpoint had been measured).
Groups:
- Total: Total of all reporting groups
Arm/Group | Nutrition With Finger-Food | Nutrition Without Finger-Food | Total
Number analyzed (Participants) | 20 | 23 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 85.3 (8.6) | 82.3 (7.6) | 83.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 20 | 23 | 43

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Measure of Ingesta
Description: Quantitative measure of ingesta (calorie and protein intake)
Time Frame: Monthly: From date of finger-food's implementation until the date of the end of the study (assessed up to 6 months)
Measure: Mean (95% Confidence Interval); unit: Kilocalories
Arm/Group | Nutrition With Finger-Food | Nutrition Without Finger-Food
Number analyzed (Participants) | 20 | 23
Kilocalories
  M-1 | 941.1 [796.5 to 1086] | 910.1 [759.8 to 1060]
  M1 | 1001 [858.8 to 1143] | 862.9 [712.6 to 1013]
  M2 | 984 [839.5 to 1129] | 843.4 [673.4 to 1013]
  M3 | 1073 [925.1 to 1220] | 865.1 [684 to 1046]
  M4 | 1065 [917.1 to 1212] | 971.9 [776.7 to 1167]
  M5 | 1055 [907.4 to 1202] | 765.9 [551.4 to 980.5]
  M6 | 1051 [900.3 to 1202] | 647.6 [366 to 929.2]
Statistical Analysis 1: Comparison: Nutrition With Finger-Food vs Nutrition Without Finger-Food; Test type: Superiority; p < 0.0001, Mixed Models Analysis

ADVERSE EVENTS:
Description: Death, serious adverse event and other (non serious adverse event) were not assessed for the study
Arm/Group | Nutrition With Finger-Food | Nutrition Without Finger-Food
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT02925728/Prot_SAP_000.pdf